CLINICAL TRIAL: NCT02652052
Title: Hematopoietic Stem Cell Transplant Survivors Study (HTSS Study)
Brief Title: Hematopoietic Stem Cell Transplant Survivors Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-004683; NCI-2021-14235 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-11-19; First posted 2016-01-11 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Stem Cell Transplant
MeSH Terms: interventions — Quercetin; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Observational (Other): Standard of Care - Observation Only
  Interventions: Other: Standard of Care - Observation Only
- Group 2: Dasatinib & Quercetin (Experimental): Interventional: The drugs dasatinib and quercetin will be used in this arm
  Interventions: Drug: Group 2: Quercetin; Drug: Group 2: Dasatinib

INTERVENTIONS:
Other: Standard of Care - Observation Only — Control Arm - Observation only
  Arms: Group 1: Observational
Drug: Group 2: Quercetin — Quercetin - take four 250mg capsules daily (total 1000 mg daily) for 3 consecutive days.
  Other Names: Quercetin
  Arms: Group 2: Dasatinib & Quercetin
Drug: Group 2: Dasatinib — Dasatinib - take one 100 mg tablet by mouth once daily for 3 consecutive days
  Other Names: Dasatinib
  Arms: Group 2: Dasatinib & Quercetin

SUMMARY:
The investigators hope to find the proof of principle concept from this pilot study so that the investigators can design a clinical trial based on the results of the explanatory hypothesis.

DETAILED DESCRIPTION:
Hematopoietic Stem Cell Transplant (HSCT) survivors are at an increased risk for premature aging. No one has evaluated the biologic markers of premature aging and senescence in HSCT survivors and their correlation with clinical outcomes, lifestyle, and nutrition. The investigators will evaluate age-related changes in HSCT survivors, with specified measures of premature aging, and employ therapeutic opportunities based on targeting senescent cells by conducting the first in-human pilot study of senolytic drugs (in HSCT survivors utilizing a combination of senolytics).

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT patients surviving ≥ 1 year post-HSCT
* Diagnosis of both malignant and non-malignant conditions as HSCT indications
* HSCT survivors receiving any type of conditioning chemo/radiotherapy for HSCT
* Ability to provide written and verbal informed consent
* Age ≥ 18 years
* Platelets > 50,000 per microliter
* Hemoglobin (HB) > 9/dL
* Absolute neutrophil count (ANC) > 1000 per microliter

Exclusion Criteria:

* HSCT survivor with human immunodeficiency virus (HIV) infection
* HSCT survivor with active hepatitis B or C HSCT survivor on any TKI for either Philadelphia chromosome positive cancers or for graft versus host disease (GVHD) treatments or for any other indication (e.g., imatinib for gastrointestinal stromal tumor [GIST], sorafenib for FLT3+ acute myeloid leukemia [AML] etc)
* HSCT survivor with any post-transplant maintenance chemotherapy
* Post-(allogeneic) transplant relapse of cancer
* Active progressive CHRONIC chronic or overlap GVHD (per the National Institute of Health [NIH] chronic GVHD criteria)
* Presence of uncontrolled psychiatric disorder
* Patient unable to give informed consent
* Extremely poor overall prognosis (<6 months as deemed by the primary transplant physician)
* HSCT survivors with confirmed drug addiction
* HSCT survivors with active coronary artery disease (CAD) [including angina] or active congestive heart failure (CHF)
* International HSCT survivors in whom loss to follow-up would be a concern as deemed by primary transplant physician
* Known hypersensitivity or allergy to dasatinib, or quercetin
* Presence of uncontrolled lupus
* Presence of uncontrolled pleural/pericardial effusions or ascites
* Presence of active new cancer (solid or hematologic) except non-melanoma skin cancers
* Presence of progeroid syndromes in family
* Invasive fungal or viral infection not responding to appropriate antifungal or antiviral therapies.
* Creatinine clearance < 60 mL/min/1.73 m2 based on the Cockcroft-Gault
* Inability to tolerate oral medications
* Presence or history of significant liver disease with total bilirubin and/or alkaline phosphatase (ALP) > 2 x upper limit normal (unless deemed to be due to Gilbert's syndrome) or as per clinical judgement
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN) or as per clinical judgement
* Active progressive ACUTE graft-versus-host disease
* Active progressive OVERLAP graft-versus-host disease
* Patients taking medications that are sensitive substrates or substrates with a narrow therapeutic range for CYP3A4, CYP2C8, CYP2C9, or CYP2D6 or strong inhibitors or inducers of CYP3A4(e.g. cyclosporine, tacrolimus or sirolimus). If antifungals are absolutely necessary from infectious disease perspective, then they will be allowed only if the levels are therapeutic. Levels will be checked at baseline and also at day +4 post intervention
* Patients taking H2-antagonists or proton pump inhibitors
* Patients on therapeutic doses of anticoagulants (e.g. warfarin, heparin, low molecular weight heparin, factor Xa inhibitors etc)
* On antiplatelet agents (e.g. full dose aspirin, clopidogrel etc.). Baby aspirin if absolutely necessary from cardiac perspective will be allowed.
* On any quinolone antibiotic therapy for treatment or for prevention of infections.
* Corrected QT (QTc) > 450 msec. Common drugs that are well known in prolonging QTc include azithromycin, citalopram, escitalopram, fluconazole, and pentamidine. Baselines electrocardiogram (EKG) will be obtained in each patient and if QTc > 450 msec, then they will be excluded from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Frailty | Up to 180 days
  Evaluate the association of frailty with measures of senescence in HSCT survivors - level of frailty as assessed by FRIED

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne R. Hayman, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials